CLINICAL TRIAL: NCT05464979
Title: Clinical Effects of Esketamine Induction Intubation Versus Conventional Induction Intubation in ICU Patients: a Single-center Randomized Clinical Trial
Brief Title: Esketamine Induction Intubation in ICU Patients.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ZJC202203
Record Dates: First submitted 2022-07-14; First posted 2022-07-19 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2022-07

CONDITIONS: Critically Ill Patients
Keywords: Esketamine; Tracheal intubation; Hemodynamics
MeSH Terms: interventions — Esketamine; Ketamine; Midazolam; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esketamine intubation group (Experimental): Esketamine at 0.5-1.0 mg/kg BW and rocuronium bromide at 0.6 mg/kg BW was given intravenously for induction intubation. After the intubation was completed, esketamine was continuously pumped at 0.3-1.5 mg/kg/h to maintain sedation. The Richmond Agitation Sedation Scale (RASS) was used to assess the sedation of patients every 1 hour and maintains a RASS score of -2 to 0.
  Interventions: Drug: Esketamine Hydrochloride 28 Mg in 0.2 mL NASAL SOLUTION [Spravato]
- Conventional intubation group (Placebo Comparator): Midazolam at 0.1mg/kg BW, fentanyl at 1ug/kg BW, rocuronium bromide at 0.6mg/kg BW was given intravenously for induction intubation; After the intubation was completed, sufentanil at 0.1 μg/kg/h was administered for analgesia, and remazolam tosylate at an initial dose of 0.075 mg/kg/h was administered for sedation, and the dose of remazolam tosylate was adjusted according to the RASS score. The RASS score was assessed every 1 h and maintained at -2 to 0.
  Interventions: Drug: midazolam, fentanyl

INTERVENTIONS:
Drug: Esketamine Hydrochloride 28 Mg in 0.2 mL NASAL SOLUTION [Spravato] — Esketamine at 0.5-1.0 mg/kg BW and rocuronium bromide at 0.6 mg/kg BW was given intravenously for induction intubation. After the intubation was completed, esketamine was continuously pumped at 0.3-1.5 mg/kg/h to maintain sedation.
  Other Names: (S)-ketamine
  Arms: Esketamine intubation group
Drug: midazolam, fentanyl — Midazolam at 0.1mg/kg BW, fentanyl at 1ug/kg BW, rocuronium bromide at 0.6mg/kg BW was given intravenously for induction intubation; After the intubation was completed, sufentanil at 0.1 μg/kg/h was administered for analgesia, and remazolam tosylate at an initial dose of 0.075 mg/kg/h was administered for sedation, and the dose of remazolam tosylate was adjusted according to the RASS score.
  Arms: Conventional intubation group

SUMMARY:
Intubation in the intensive care unit (ICU) is usually an emergency. Pathophysiological changes such as shock, respiratory failure, and metabolic acidosis in critically ill patients can significantly increase the incidence of adverse events during intubation.

Studies have shown that esketamine has no significant effect on body metabolism, endocrine system, liver, kidney, intestinal function and coagulation function. In terms of drug metabolism, esketamine has high bioavailability, short half-life, faster and more comfortable recovery of patients, and not only has the advantage of providing stable hemodynamics during endotracheal intubation, but also counteracts the respiratory depression caused by opioids. In addition, esketamine has antidepressant and anti-inflammatory properties. The investigators also found that combined prophylactic and therapeutic use of esketamine could attenuate systemic inflammation and inflammatory multi-organ injury in mice after CLP-induced lethal sepsis.

This project aims to study the clinical effect of esketamine induction intubation and conventional induction intubation in ICU patients.

DETAILED DESCRIPTION:
Esketamine is the S-enantiomer of ketamine and has been approved for clinical use by the National Medical Products Administration (NMPA) in 2019. Studies have shown that esketamine has no significant effect on metabolism, endocrine system, liver, kidney, intestinal function and coagulation function. It is mainly used in combination with sedatives (such as propofol, etc.) or alone to induce and implement general anesthesia. The phase III clinical study on the application of esketamine in the induction and maintenance of general anesthesia in laparoscopic surgery showed that the recovery time of the esketamine group was significantly shorter than that of the ketamine group when the same clinical anesthesia effect was achieved. Esketamine has the effect of dissociative anesthesia, which can maintain better spontaneous breathing of patients while satisfying outpatient examinations or operations, and this feature helps maintain circulatory stability, especially in patients with shock. Esketamine has sympathomimetic properties. In patients with potentially unstable cardiac disease (eg, septic cardiomyopathy), esketamine is the preferred choice for induction of anesthesia, especially in combination with midazolam. Esketamine is also the preferred choice for anesthesia induction in patients with bronchospasm, which can protect patients from bronchospasm during induction.

Studies have found that esketamine has antidepressant and anti-inflammatory effects in addition to its analgesic, sedative and anesthetic effects. Clinical studies have shown that esketamine (0.25 mg/kg, 40 min infusion time) can rapidly improve the depressive symptoms of patients with treatment-resistant depression. The antidepressant effects of esketamine may be closely related to its anti-inflammatory effect. During cardiopulmonary bypass surgery, anesthesia induction was supplemented with 1-3 mg/kg esketamine, anesthesia maintenance was supplemented with 2-3 mg/kg/h esketamine, anesthesia maintenance time was 283 minutes, the total amount of esketamine was 1580mg on average. Esketamine decreased plasma levels of IL-6 (6 h after opening the aorta) and IL-8 (1 and 6 h after opening the aorta) and increased plasma levels of IL-10 (1 h after opening the aorta). In the investigators' preliminary study on the role of esketamine in systemic inflammation induced by lipopolysaccharide (LPS), the investigators found that in systemic LPS (5 mg/kg)-induced systemic inflammation model, esketamine (10 mg/kg, IP) was administrated twice 24 hours before LPS administration and 10 minutes after LPS administration. The plasma levels of IL-6, IL-17A and interferon γ (IFN-γ) were significantly decreased 24 h after LPS administration in mice. However, the efficacy and safety of esketamine for tracheal intubation in ICU patients is still unclear, and no relevant clinical studies have been reported.

The investigators will include adult patients subjected to tracheal intubation in the ICU strictly according to the inclusion and exclusion criteria to investigate the efficacy and safety of esketamine for tracheal intubation in ICU patients.

Enrolled patients were randomly assigned to two groups: the esketamine intubation group and the conventional intubation group. In esketamine intubation group, esketamine at 0.5-1.0 mg/kg BW and rocuronium bromide at 0.6 mg/kg BW was given intravenously for induction intubation. After the intubation was completed, esketamine was continuously pumped at 0.3-1.5 mg/kg/h to maintain sedation. In conventional intubation group, Midazolam at 0.1mg/kg BW, fentanyl at 1ug/kg BW, rocuronium bromide at 0.6mg/kg BW was given intravenously for induction intubation; After the intubation was completed, sufentanil at 0.1 μg/kg/h was administered for analgesia, and remazolam tosylate at an initial dose of 0.075 mg/kg/h was administered for sedation, and the dose of remazolam tosylate was adjusted according to the RASS score.

Five tubes of venous blood were collected and sent to the laboratory and immunology department of Union Hospital affiliated to Tongji Medical College, Huazhong University of Science and Technology, before intubation and 1, 2, 3 and 7 days after intubation, and five tests including blood routine, coagulation, liver function, kidney function, electrolytes, C-reactive protein, myocardial enzyme, BNP, lymphocyte subsets and cytokines were performed. A tube of arterial blood was collected before intubation and 1, 2, 3 and 7 days after intubation to detect arterial blood gas in the ICU.

If the adverse events of esketamine appear during the study, patients or authorized client withdraw from the study actively, or drugs that seriously affect systemic inflammation and immune function (such as non-steroidal anti-inflammatory drugs, immunosuppressants, immunoenhancers, high doses of hormones (more than 10mg prednisolone per day or equivalent dose of other hormones, etc.) were used in clinical treatment, the study will be terminated. In this study, adverse reactions were evaluated daily after inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years old without restriction of gender, race, religion, creed or nationality;
* No sedative drugs with elimination half-life were used before inclusion in the study;
* Patients and/or their family members know and agree to participate in the trial.

Exclusion Criteria:

* Allergic to esketamine or midazolam;
* Patients with cardiac arrest during intubation;
* Patients with suspected increased intracranial pressure;
* bradycardia (heart rate below 50 beats/min) or atrioventricular block;
* Untreated or undertreated patients with hyperthyroidism;
* Diseases that may affect immune-related indicators, including autoimmune diseases (rheumatoid arthritis and systemic lupus erythematosus, etc.), and malignant hematological tumours (leukaemia and lymphoma, etc.);
* Received radiotherapy or chemotherapy or received immunosuppressive drug treatment within the past 30 days, or received more than 10 mg of prednisolone per day (or other hormones at the same dose) continuous treatment;
* History of solid organ or bone marrow transplantation;
* Chronic nephrosis;
* Severe chronic liver disease (child-Pugh: Grade C);
* alcohol or opioid dependence, mental illness, or severe cognitive impairment;
* Pregnant or breastfeeding;
* Patients and/or their family members refuse to participate in the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Level of systolic blood pressure, diastolic blood pressure and mean arterial pressure | 5 minutes before induction
  Systolic blood pressure, diastolic blood pressure and mean arterial pressure
Level of systolic blood pressure, diastolic blood pressure and mean arterial pressure | 0 hour after induction
  Systolic blood pressure, diastolic blood pressure and mean arterial pressure
Level of systolic blood pressure, diastolic blood pressure and mean arterial pressure | 0 hour after intubation
  Systolic blood pressure, diastolic blood pressure and mean arterial pressure
Level of systolic blood pressure, diastolic blood pressure and mean arterial pressure | 1 minute after intubation
  Systolic blood pressure, diastolic blood pressure and mean arterial pressure
Level of systolic blood pressure, diastolic blood pressure and mean arterial pressure | 5 minutes after intubation
  Systolic blood pressure, diastolic blood pressure and mean arterial pressure
Level of systolic blood pressure, diastolic blood pressure and mean arterial pressure | 10 minutes after intubation
  Systolic blood pressure, diastolic blood pressure and mean arterial pressure
Level of systolic blood pressure, diastolic blood pressure and mean arterial pressure | 30 minutes after intubation
  Systolic blood pressure, diastolic blood pressure and mean arterial pressure
Level of systolic blood pressure, diastolic blood pressure and mean arterial pressure | 60 minutes after intubation
  Systolic blood pressure, diastolic blood pressure and mean arterial pressure
Level of heart rate and respiratory rate | 5 minutes before induction
  Heart rate and respiratory rate
Level of heart rate and respiratory rate | 0 hour after induction
  Heart rate and respiratory rate
Level of heart rate and respiratory rate | 0 hour after intubation
  Heart rate and respiratory rate
Level of heart rate and respiratory rate | 1 minute after intubation
  Heart rate and respiratory rate
Level of heart rate and respiratory rate | 5 minutes after intubation
  Heart rate and respiratory rate
Level of heart rate and respiratory rate | 10 minutes after intubation
  Heart rate and respiratory rate
Level of heart rate and respiratory rate | 30 minutes after intubation
  Heart rate and respiratory rate
Level of heart rate and respiratory rate | 60 minutes after intubation
  Heart rate and respiratory rate
Level of pulse oximetry | 5 minutes before induction
  Pulse oximetry
Level of pulse oximetry | 0 hour after induction
  Pulse oximetry
Level of pulse oximetry | 0 hour after intubation
  Pulse oximetry
Level of pulse oximetry | 1 minute after intubation
  Pulse oximetry
Level of pulse oximetry | 5 minutes after intubation
  Pulse oximetry
Level of pulse oximetry | 10 minutes after intubation
  Pulse oximetry
Level of pulse oximetry | 30 minutes after intubation
  Pulse oximetry
Level of pulse oximetry | 60 minutes after intubation
  Pulse oximetry

SECONDARY OUTCOMES:
Doses of epinephrine and norepinephrine | At 1 hour after intubation
  Epinephrine and norepinephrine doses
Doses of epinephrine and norepinephrine | At 24 hours after intubation
  Epinephrine and norepinephrine doses
Plasma cytokine levels | On day 3 after intubation
  IL-2、IL-4、IL-6、IL-10、IL-17A、IFN-γ、TNF-α
Acute physiology and chronic health evaluation (APACHE) Ⅱ score | 0 hour after study inclusion
  0-67, higher scores correspond to more severe disease and a higher risk of death
Acute physiology and chronic health evaluation (APACHE) Ⅱ score | 1 day after intubation
  0-67, higher scores correspond to more severe disease and a higher risk of death
Acute physiology and chronic health evaluation (APACHE) Ⅱ score | 2 days after intubation
  0-67, higher scores correspond to more severe disease and a higher risk of death
Acute physiology and chronic health evaluation (APACHE) Ⅱ score | 3 days after intubation
  0-67, higher scores correspond to more severe disease and a higher risk of death
Acute physiology and chronic health evaluation (APACHE) Ⅱ score | 7 days after intubation
  0-67, higher scores correspond to more severe disease and a higher risk of death
Sequential organ failure assessment (SOFA) score | 0 hour after study inclusion
  0-43, higher scores correspond to more severe disease
Sequential organ failure assessment (SOFA) score | 1 day after intubation
  0-43, higher scores correspond to more severe disease
Sequential organ failure assessment (SOFA) score | 2 days after intubation
  0-43, higher scores correspond to more severe disease
Sequential organ failure assessment (SOFA) score | 3 days after intubation
  0-43, higher scores correspond to more severe disease
Sequential organ failure assessment (SOFA) score | 7 days after intubation
  0-43, higher scores correspond to more severe disease
Hamilton Anxiety Scale (HAMA) Score | 1 day after extubation
  0-29，higher scores correspond to more severe anxiety
Hamilton Depression Scale (HAMD) Score | 1 day after extubation
  0-35，higher scores correspond to more severe depression
The number of intubation attempts | At intubation procedure
  Intubation times
Mechanical ventilation-free time | 7 days of after inclusion
  Time to weaning from invasive mechanical ventilation
28-day ICU and in-hospital mortality | Up to 28 days after inclusion
  Death within 28 days after hospitalization or ICU stay
90-day readmission rates | Up to 90 days after discharge from hospital
  Hospitalized again within 90 days after discharge from hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Jiancheng Zhang, MD, PhD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Department of Critical Care Medicine, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
After publication, the data supporting the findings of this study can be provided by the corresponding author upon reasonable request. Participant data without names and identifiers can be provided by the corresponding author and the Wuhan Union Hospital after approval. The research team will provide an email address for communication purposes once approval is obtained regarding sharing the data with others. The proposal with detailed description of the study objectives and statistical analysis plan will be needed for evaluation of the purpose for the data request. Additional materials may also be required during the process of evaluation.
Supporting Information: Study Protocol
Time Frame: Six months after publication.
Access Criteria: Upon reasonable request.

REFERENCES:
- [Derived] Zhang X, Zhao X, Xu J, Liu H, Yuan S, Zhang J. Efficacy and safety of esketamine for emergency endotracheal intubation in ICU patients: a double-blind, randomized controlled clinical trial. Sci Rep. 2025 Feb 19;15(1):6089. doi: 10.1038/s41598-025-91016-w. PMID 39972022